CLINICAL TRIAL: NCT00317083
Title: Effect of Obstructive Sleep Apnea Syndrome Associated With Obesity on Cough Reflex Threshold to Citric Acid
Brief Title: Cough Reflex and Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bichat Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: JG-2006-BCH
Record Dates: First submitted 2006-04-17; First posted 2006-04-24 (Estimated); Last update posted 2006-04-24 (Estimated); Status verified 2004-01

CONDITIONS: Sleep Apnea Syndrome
Keywords: Cough Reflex; Citric acid; Obesity; Sleep apnea syndrome
MeSH Terms: conditions — Sleep Apnea Syndromes; Obesity

INTERVENTIONS:
Procedure: Cough reflex test

SUMMARY:
Up to 70% of obese patients undergoing bariatric surgery have obstructive sleep apnea syndrome (OSAS). OSAS is responsible for laryngeal sensory impairment. As the afferent neural pathway involved in the initiation of cough is located in the laryngeal epithelium, cough reflex sensitivity may be decreased in obese OSAS patients. The researchers therefore conducted this study to determine the effect of OSAS associated with obesity on cough reflex sensitivity, assessed by cough reflex threshold to an inhaled irritant (citric acid).

DETAILED DESCRIPTION:
Obese patients undergoing scheduled bariatric surgery underwent a cough challenge as part of their routine preoperative evaluation. Patients were classified as presenting OSAS if apnea-hypopnea index obtained from preoperative full-night polysomnography was greater than 5/hour. Cough threshold was measured with citric acid. Increasing concentrations of mouth- nebulized citric acid (2.5, 5, 10, 20, 40, 80, 160, 320 and 640 mg/mL) were delivered during inspiration until a cough was elicited. The citric acid concentration eliciting one cough (C1) was defined as the cough reflex threshold.

ELIGIBILITY:
Inclusion Criteria:

* Obese patient scheduled to undergo bariatric surgery

Exclusion Criteria:

* Age less than 18
* Active smoking
* Psychotropic medication
* Angiotensin-converting enzyme inhibitor or angiotensin II receptor antagonist medication
* Pregnancy
* Anesthesia or endotracheal intubation during the previous month
* Allergic rhinitis
* Upper airway or bronchopulmonary infection during the previous month
* Chronic cough
* Chronic respiratory disease
* Pharyngolaryngeal disease
* Neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2001-11; Study Completion 2003-02

PRIMARY OUTCOMES:
To compare cough reflex threshold to citric acid between obese OSAS patients and obese non-OSAS patients

SECONDARY OUTCOMES:
To correlate OSAS severity assessed by apnea-hypopnea index and cough reflex threshold to citric acid

CONTACTS AND LOCATIONS:
Overall Officials: Jean Guglielminotti, Principal Investigator — Anesthesiology Department, Bichat Hospital
Locations (1):
- Anesthesiology Department, Bichat Hospital, Paris, France

REFERENCES:
- [Background] Nguyen AT, Jobin V, Payne R, Beauregard J, Naor N, Kimoff RJ. Laryngeal and velopharyngeal sensory impairment in obstructive sleep apnea. Sleep. 2005 May;28(5):585-93. doi: 10.1093/sleep/28.5.585. PMID 16171271